CLINICAL TRIAL: NCT00600080
Title: The Comparative Clinical Performance of the Etafilcon A Lens and the DAILIES AquaComfort Plus Lens
Brief Title: A Comparison of Two Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0729
Record Dates: First submitted 2007-12-21; First posted 2008-01-24 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- etafilcon A first nelfilcon A second (Other): etafilcon A worn daily during week 1, nelfilcon A worn daily for week 2
  Interventions: Device: etafilcon A; Device: nelfilcon A
- nelfilcon A first, etafilcon A second (Other): nelfilcon A worn daily during week 1, etafilcon A worn daily for week 2
  Interventions: Device: etafilcon A; Device: nelfilcon A

INTERVENTIONS:
Device: etafilcon A — contact lens worn daily for one week (first or second week depending on arm)
  Other Names: 1-DAY ACUVUE MOIST
Device: nelfilcon A — Contact lens worn daily for one week (first or second week depending on arm)
  Other Names: DAILIES AquaComfort Plus

SUMMARY:
This study seeks to evaluate the clinical performance of a recently improved daily disposable contact lens to an established daily disposable contact lens that contains a wetting agent.

ELIGIBILITY:
Inclusion Criteria:

1. They are of legal age (18 years) and capacity to volunteer.
2. They understand their rights as a research subject and are willing to sign a Statement of Informed Consent.
3. They are willing and able to follow the protocol.
4. They would be expected to attain at least 6/9 (20/30) in each eye with the study lenses.
5. They are able to wear contact lenses with a back vertex power of -1.00 to -6.00DS.
6. They have a maximum of 1.00D of refractive astigmatism (i.e. ≤ 1.00 DC).
7. They have successfully worn contact lenses within six months of starting the study. -

Exclusion Criteria:

1. They have an ocular disorder which would normally contra-indicate contact lens wear.
2. They have a systemic disorder which would normally contra-indicate contact lens wear.
3. They are using any topical medication such as eye drops or ointment.
4. They are aphakic.
5. They have had corneal refractive surgery.
6. They have any corneal distortion resulting from previous hard or rigid lens wear or has keratoconus.
7. They are pregnant or lactating.
8. They have grade 2 or greater of any of the following ocular surface signs: corneal oedema, corneal vascularisation, corneal staining, tarsal conjunctival changes or any other abnormality which would normally contraindicate contact lens wear.
9. They have any infectious disease (e.g. hepatitis) or any immunosuppressive disease (e.g. HIV).
10. They have diabetes.
11. They have taken part in any other clinical trial or research, within two weeks prior to starting this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eurolens Research, The University of Manchester Dpt. of Optometry & Neuroscience, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty subjects were enrolled onto the study to wear contact lenses for two weeks on a daily wear basis.
Pre-assignment Details: Sixty subjects enrolled and sixty subjects completed.
Groups:
- Etafilcon A/Nelfilcon A: etafilcon A worn daily during week 1, nelfilcon A worn daily for week 2.
- Nelfilcon A/Etafilcon A: nelfilcon A worn daily during week 1, etafilcon A worn daily for week 2.
Period: Period 1: Baseline to One-week
Arm/Group | Etafilcon A/Nelfilcon A | Nelfilcon A/Etafilcon A
Started | 28 | 32
Completed | 28 | 32
Not Completed | 0 | 0
Period: Period 2: One-week to Two-weeks
Arm/Group | Etafilcon A/Nelfilcon A | Nelfilcon A/Etafilcon A
Started | 28 (This is a crossover study, arms are switched at period change.) | 32 (This is a crossover study, arms are switched at period change.)
Completed | 28 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects are those who were enrolled and randomized to a study arm. Sixty subjects were enrolled and sixty subjects completed.
Groups:
- All Subjects: All subjects crossed over to use each treatment for one week
Arm/Group | All Subjects
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 17
Region of Enrollment [Number; unit: participants]
  United Kingdom | 60

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Measured using high contrast and low contrast vision charts without the use of spectacles (glasses) or refraction equipment (for contact lens wearers). Values are on the logMar scale where lower values (< 0) refer to 'better' values of sight. These scores are converted from a Snellen eye chart examination.
Time Frame: 2-week
Population: Subjects analyzed are those who were enrolled, randomized to a study arm, and completed the study.
Measure: Mean (Standard Deviation); unit: logMAR scale
Groups:
- Nelfilcon A: All subjects who wore nelfilcon A lenses for one week
- Etafilcon A: All subjects who wore etafilcon A lenses for one week
Arm/Group | Nelfilcon A | Etafilcon A
Number analyzed (Participants) | 60 | 60
logMAR scale
  High Contrast | -0.10 (0.07) | -0.10 (0.07)
  Low Contrast | 0.17 (0.09) | 0.18 (0.09)

2. Secondary Outcome: Subject-reported Overall Product Performance
Description: Subjects were asked to rate lens performance on a scale of 0 to 100 point scale (0= "Extremely poor" or "Cannot use lenses" and 100= "Excellent" or "Highly impressed with these lenses overall"). The average score is reported. A factor analysis was used to identify the questions pertaining to product performance, a factor loading of 0.4 or greater was used.
Time Frame: 2-week
Population: Analyzed subjects were those who were enrolled and randomized to a study arm.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Nelfilcon A | Etafilcon A
Number analyzed (Participants) | 60 | 60
units on a scale | 86.5 (11.3) | 87.7 (12.3)

3. Secondary Outcome: Optimum Lens Fit
Description: Number of subjects that measured as an optimum fit. Lens fit will be assessed using the following evaluations: horizontal and vertical centration, corneal coverage and movement. Normally, for an acceptable fit, centration and movement will fall within currently accepted clinical criteria [between -1 and +1 on a -2 to +2 grading scale.
Time Frame: Baseline, 1-week, 2-week
Population: Subjects analyzed were those who were enrolled, randomized to a study arm, and completed the study.
Measure: Number; unit: participants
Arm/Group | Nelfilcon A | Etafilcon A
Number analyzed (Participants) | 60 | 60
participants
  At Dispensing | 22 | 18
  At Follow-up | 18 | 18

4. Primary Outcome: Subjective Lens Comfort
Description: as for outcome 2
Time Frame: 2-week
Population: Subjects analyzed were those who were enrolled, randomized to a study arm, and completed the study.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nelfilcon A | Etafilcon A
Number analyzed (Participants) | 60 | 60
units on a scale | 86.0 (13.9) | 88.2 (12.4)

ADVERSE EVENTS:
Groups:
- Nelfilcon A First Etafilcon A Second: nelfilcon A worn daily during week 1, etafilcon A worn daily for week 2
Arm/Group | Etafilcon A First Nelfilcon A Second | Nelfilcon A First Etafilcon A Second
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication requires agreement and written authorization from Sponsor.